CLINICAL TRIAL: NCT03291535
Title: Virtual Hypertension Management Pilot: Randomized Evaluation of Electronic Health Record-connected Blood Pressure Cuffs in a Clinical Pharmacist Panel.
Brief Title: Virtual Hypertension Management Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, N. Lance Downing, MD, Clinical Assistant Professor of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 12397
Record Dates: First submitted 2017-08-17; First posted 2017-09-25 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Hypertension; Electronic Health Record; Digital Health
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): This arm will consist of the usual care of management of hypertension by a clinical pharmacist.
  Interventions: Other: Usual care
- Intervention (Active Comparator): This arm will consistent of usual care plus the addition of a blood pressure cuff that will allow patients to upload data to the electronic health record via a secure portal.
  Interventions: Other: Connected-device

INTERVENTIONS:
Other: Connected-device — This intervention will allow patients to upload blood pressure data automatically from a blood pressure cuff into the electronic health record.
  Arms: Intervention
Other: Usual care — This intervention will consist of usual clinical care as determined by the clinical pharmacist.
  Arms: Control

SUMMARY:
Investigators are examining the quality improvement impact of providing patients with a an electronic health record-connected blood pressure cuff. Investigators will give half of patients already eligible for hypertension management within a clinical pharmacist panel, the ability to upload their blood pressure data into Stanford's electronic health record.

ELIGIBILITY:
Inclusion Criteria:

* Hypertension as defined by clinical pharmacist usual care panel (2 or more readings of blood pressure >140/90)

Exclusion Criteria:

* Pregnancy
* Chronic kidney disease III or IV
* Systolic heart failure with ejection fraction <35%
* Current use of 3 or more anti-hypertension drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure over time in control group vs. the intervention group | From enrollment to 6 months later
  Difference in the change in blood pressure between the control group and intervention group.

SECONDARY OUTCOMES:
Patient visits | From enrollment to 6 months later
  Measurement of the number of in-person visits
Patient remote interactions | From enrollment to 6 months later
  Measurement of the number of patient phone calls plus patient-portal messages to the clinical pharmacist
Medication changes | From enrollment to 6 months later
  Number of changes in medication or medication dose
Blood pressure control | From enrollment to 6 months later
  Time to reach target blood pressure control (Adults 18-59 years of age <140/90 mm Hg, Adults 60-85 years of age, without a diagnosis of diabetes, <150/90 mm Hg, Adults 60-85 years of age, with a diagnosis of diabetes, <140/90 mm Hg)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Stanford Primary Care, Portola Valley, California
  - Stanford Primary Care Clinic, Santa Clara, California

IPD SHARING:
Plan to Share IPD: Undecided
Undecided, this is a quality improvement project.